CLINICAL TRIAL: NCT00173576
Title: Clinical Study of SARS in Children
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9461700732; NSC92-2751-B-002-013-Y
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-10-27 (Estimated); Status verified 2005-08

CONDITIONS: Epidemiology

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Severe acute Respiratory Syndrome (SARS) is an emerging infectious disease. It is caused by a novel SARS-associated coronavirus. According to the epidemiological data, it is highly infectious by intimate contact, respiratory secretion, or direct contact with infectious body fluid. By June 1, 2003, Center for Disease Control Taiwan, R.O.C reported 677 probable SARS cases. Among them, 93.2% (631/677) were more than 20 years old. Only 6.8% (46/677) were under 20 years old. Usually the major hosts of respiratory viruses are children, but evidence up to now shows that SARS is mainly a disease of adults. The data of clinical presentation and epidemiological prevalence in teenage group and children are lacking. Therefore, this project is aimed at the children and teenager among 1 month to eighteen years old. Seroepidemiology of SARS-CoV infection in children would be investigated. Patients who admitted to pediatric wards or visited ER and received blood sampling due to the need of clinical diagnosis/management would be enrolled. After the necessary laboratory examinations were done, the remaining serum would be collected and tested for anti-SARS-CoV IgG by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 1 month to 18 years old
* Received blood sampling during admission or at emergency department due to the need of clinical diagnosis/management

Exclusion Criteria:

-

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800
Dates: Start 2003-04; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, MD, PhD, Principal Investigator — Department of Pediatrics, College of Medicine, National Taiwan University and Graduate Institute of Preventive Medicine, College of Public Health, National Taiwan University